CLINICAL TRIAL: NCT04555148
Title: A Prospective, Open-label, Randomized, Multi-center, Phase 2a Study to Evaluation the Dose Response, Efficacy and Safety of Hyper-Ig (Hyper-immunoglobulin) GC5131 in Patients With COVID-19
Brief Title: COVIDIG (COVID-19 Hyper-ImmunoGlobulin)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GC5131A-HIG_P0201
Record Dates: First submitted 2020-09-16; First posted 2020-09-18 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Saline
  Interventions: Other: Placebo
- Low dose Treatment (Experimental): Low dose treatment
  Interventions: Biological: GC5131
- Medium dose Treatment (Experimental): Medium dose Treatment
  Interventions: Biological: GC5131
- High dose Treatment (Experimental): High dose Treatment
  Interventions: Biological: GC5131

INTERVENTIONS:
Biological: GC5131 — COVID19 Hyper-Immunoglobulin
  Arms: High dose Treatment; Low dose Treatment; Medium dose Treatment
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of 5131A for hospitalized patients of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* The COVID-19 patient who diagnosed by PCR within 3 days prior to randomized And who is hospitalized with COVID-19 related symptoms
* The subject who has symptoms of COVID-19 within 7 days
* The subject with pneumonia confirmed by imaging diagnosis related to COVID-19 OR a 70-year-old or older OR 60-year-old or older with underlying disease (diabetes or hypertension or obesity or smoker)
* Willing and able to provide written informed consent prior to performing study procedures

Exclusion Criteria:

* asymptomatic patient
* The subject who requiring mechanical ventilation or ECMO
* The subject who are underlying oxygen therapy before affected by COVID-19
* The subject who have received antiviral drugs for other disease within 4 weeks
* History of allergy to IVIG or plasma products
* The subject who received IVIG or convalescent plasma from a person who recovered from COVID-19
* IgA deficiency
* Cretinine > 2 X ULN
* The subject with a history of thrombosis or high risk of thromboembolism
* The subject with reduced heart function [NYHA (New York Heart Association) Functional Class III or IV]; or cerebral cardiovascular disorder or a patient with the medical history (ischemic disease, cardiovascular disease, cerebrovascular disorder, blood vessel disorder, etc.)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-09-19 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Ordinal scale outcome | 7, 14, 21, 28 days
  The percent of participants changed by 2 points or more

SECONDARY OUTCOMES:
Viral negative | 1, 3, 5, 7, 10 days
  The percents of negative patients for COVID-19 virus
Change in NEWS2 (National Early Warning Score 2) | 7, 14, 21, 28 days
  The change of National Early Warning Score 2 (NEWS) from baseline
mortality | 28 days
  The percent of participants

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea